CLINICAL TRIAL: NCT06785246
Title: Grasshopper: a Novel Clinical Dashboard for Radiologists
Acronym: Grasshopper
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Principal Investigator, Jason D. Balkman, Principal Investigator, Kaiser Permanente
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 2142507
Record Dates: First submitted 2025-01-07; First posted 2025-01-21 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2025-01

CONDITIONS: Chest Infection; Pulmonary Edema - Acute
Keywords: AI; Emergency Department; Radiology; Imaging
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Intervention Model Description: Stepped wedge cluster randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Grasshopper CXR Dashboard (Experimental): Grasshopper CXR Dashboard
  Interventions: Other: Grasshopper dashboard

INTERVENTIONS:
Other: Grasshopper dashboard — Computer dashboard application for radiologists that displays relevant clinical information directly from the medical record

SUMMARY:
Does a radiology clinical dashboard increase radiologist use of specific reporting language for chest X-rays (CXRs) and thereby decrease rates of unnecessary Emergency Department (ED) prescriptions and follow-up imaging?

DETAILED DESCRIPTION:
Chest X-rays (CXR) are the most common radiologic exam, comprising nearly one third of total KPNC imaging volume. Despite high CXR utilization, diagnostic yield is frequently low, partly due to the paucity of clinical information provided to radiologists at the time of CXR interpretation, resulting in frequent nonspecific CXR assessments which include terms like "opacities" instead of diagnostic terms such as "pulmonary edema" or "pneumonia". This may contribute to over-treatment and unnecessary follow-up CT imaging. This study proposes the production deployment, active promotion, and evaluation of an innovative clinical dashboard called Grasshopper for radiologists to provide pertinent clinical information at the time of CXR interpretation. The dashboard leverages the electronic medical record to programmatically retrieve, and display select clinical notes, patient lab values, and vital signs. The Grasshopper study aims to prospectively evaluate the impact of Grasshopper on CXR report specificity in ED settings across 15 KPNC service areas, and on downstream care process measures such as prescription and imaging utilization.

ELIGIBILITY:
Kaiser Permanente Northern California CXR is ordered during emergency room visit or inpatient hospitalization

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100000 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Diagnostic CXR Reports | Through study completion, an average of 18 months.
  Number of CXR reports that employ diagnostic terms in the report impression (e.g. "negative", "pneumonia", "pulmonary edema"), compared with baseline standard of care report impressions.

SECONDARY OUTCOMES:
Number of Prescriptions after Stat CXR | Through study completion, at an average of 18 months.
  Number of antibiotic and diuretic prescriptions the patient receives after having undergone a stat CXR, compared with baseline standard of care.
Number of CT Imaging exams after Stat CXR | Through study completion, at an average of 18 months.
  Number of follow-up CT imaging exams that a patient receives after having undergone a stat CXR, compared with baseline standard of care.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaiser Permanente Northern California Division of Research, Pleasanton, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Pending further organizational guidance